CLINICAL TRIAL: NCT03271229
Title: A Randomized, Single-Blinded, Controlled Trial Comparing Conventional Platelet Rich Plasma (PRP) to Concentrated Bone Marrow Aspirate (BMAC) for Osteoarthritis of the Knee
Brief Title: Conventional Platelet-Rich Plasma Versus Concentrated Bone Marrow Stem Cell Injections for Osteoarthritis of the Knee
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shane A. Shapiro, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-008718
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Osteo Arthritis Knee
Keywords: Platelet rich plasma; bone marrow; stem cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stem Cells (Active Comparator): Participants will have Concentrated Bone Marrow Aspirate (BMAC) injections into symptomatic knee
  Interventions: Biological: Concentrated Bone Marrow Aspirate (BMAC)
- Plasma (Active Comparator): Participants will have Platelet-Rich Plasma (PRP) injections into symptomatic knee
  Interventions: Biological: Platelet-Rich Plasma (PRP)

INTERVENTIONS:
Biological: Concentrated Bone Marrow Aspirate (BMAC) — Participants will have a knee injected with BMAC stem cells harvested from the iliac crest
  Arms: Stem Cells
Biological: Platelet-Rich Plasma (PRP) — Participants will have a knee injected with Platelet-Rich Plasma (PRP) obtained from a venous whole blood draw from the antecubital vein.
  Arms: Plasma

SUMMARY:
Previous clinical trials have demonstrated the human body's own healing and regenerative cells can relieve the pain of arthritis. Bone marrow contains stem cells which can change into cells of various different tissue types, while platelet rich plasma contains growth factors. Both techniques have been shown to relieve pain and with this study the Investigators wish to compare the two treatments.

DETAILED DESCRIPTION:
Participants will be randomized into two groups. Concentrated Bone Marrow Aspirate (BMAC) or Platelet-Rich Plasma (PRP). BMAC subjects will have bone marrow aspirated from the subjects iliac crests and the cellular rich portion will be concentrated and subsequently injected into the subjects' symptomatic knee. BMAC patients will also have a venous whole blood drawn from the antecubital vein to simulate a PRP procedure. PRP subjects will have the same venous blood draw from the antecubital vein with subsequent platelet concentration. The resulting PRP will be injected into the symptomatic knee. PRP subjects will also undergo a bone marrow aspiration from the iliac crest to simulate the BMAC procedure. Follow-up at 1 week, 6 weeks, 6 months, and 12 months after injection, with repeat radiographs at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have bilateral OA and pain in one knee.
* Osteoarthritis may be primary or secondary. Knees must have Kellgren-Lawrence Grades 1-3.
* Subjects must have previously tried 6 weeks of one of the following conservative treatments: Activity modification, weight loss, physical therapy, anti-inflammatory, or injection therapy.
* Patients must be able to provide written informed consent after the nature of the study is fully explained.

Exclusion Criteria:

* Patients with abnormal hematology, serum chemistry, or screening laboratory results.
* Patients taking anti-inflammatory medications (prescription or over-the-counter), including herbal therapies, within 14 days of baseline visit.
* Patients taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within the 3 months prior to study entry.
* Patients receiving injections to the treated knee within 3 months prior to study entry.
* Patients who are pregnant or currently breast-feeding.
* Patients with systemic, rheumatic, or inflammatory disease of the knee or chondrocalcinosis, hemochromatosis, inflammatory arthritis, arthropathy of the knee associated with juxta-articular Paget's disease of the femur or tibia, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's knee joint, villonodular synovitis, and synovial chondromatosis.
* Patients with ongoing known infectious disease.
* Patients with clinically significant cardiovascular, renal, hepatic, endocrine disease, or cancer.
* Patients participating in a study of an experimental drug or medical device within 30 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Adverse Events | approximately 12 months
  The number of adverse events
Morbidity | approximately 12 months
  The number of deceased participants

CONTACTS AND LOCATIONS:
Overall Officials: Shane A Shapiro, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials